CLINICAL TRIAL: NCT06683924
Title: Comparison of Pulsed Radiofrequency Ablation and Steroid Injections of The Lateral Femoral Cutaneous Nerve for The Treatment of Meralgia Paresthetica
Brief Title: Pulsed Radiofrequency Ablation and Steroid Injections for the Treatment of Meralgia Paresthetica
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Ayşe Merve Ata, MD, Principal Investigator, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TABED 1-24-218
Record Dates: First submitted 2024-11-09; First posted 2024-11-12 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2024-11

CONDITIONS: Meralgia Paresthetica
Keywords: meralgia paresthetica; pulsed radiofrequency ablation; lateral femoral cutaneous nerve
MeSH Terms: conditions — Femoral Neuropathy | interventions — Steroids; Dexamethasone; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulsed Radiofrequency Ablation (Active Comparator): The area where the lateral femoral cutaneous nerve is seen with US will be anesthetized with 1 ml of 1% lidocaine and a 22 Gauge, 10 cm-5 mm RF cannula will be inserted. Sensory fibers will be stimulated with 0.3-0.5 V. Then, motor fibers will be stimulated up to 1.5 V. If no motor contraction is seen, LFCN will be ablated at 42 degrees Celsius for 240 seconds. The procedure will be completed with the injection of 2 ml of 2% lidocaine and 2 ml (8 mg) dexamethasone through the RF cannula.
- Steroid Injection (Active Comparator): Where the lateral femoral cutaneous nerve is visible with US, 2 ml of 2% lidocaine and 2 ml (8 mg) dexamethasone will be injected.
  Interventions: Drug: Steroid (dexamethasone) Injection

INTERVENTIONS:
Procedure: Pulsed Radiofrequency Ablation — The area where the lateral femoral cutaneous nerve is seen with US will be anesthetized with 1 ml of 1% lidocaine and a 22 Gauge, 10 cm-5 mm RF cannula will be inserted. Sensory fibers will be stimulated with 0.3-0.5 V. Then, motor fibers will be stimulated up to 1.5 V. If no motor contraction is seen, LFCN will be ablated at 42 degrees Celsius for 240 seconds. The procedure will be completed with the injection of 2 ml of 2% lidocaine and 2 ml (8 mg) dexamethasone through the RF cannula.
Drug: Steroid (dexamethasone) Injection — Where the lateral femoral cutaneous nerve is visible with US, 2 ml of 2% lidocaine and 2 ml (8 mg) dexamethasone will be injected.
  Arms: Steroid Injection

SUMMARY:
Meralgia Paresthetica (MP) is a mononeuropathy of the lateral femoral cutaneous nerve (LFCN), characterized by pain, numbness, hyperesthesia, or hypoesthesia, especially in the anterolateral thigh where the nerve has a sensory distribution. TheLFCN passes between the psoas and quadratus lumborum muscles in the iliac fossa and enters the thigh under the inguinal ligament by passing through the anterior superior iliac spine over the iliacus muscle. It superficially spreads over the sartorius muscle and receives sensation in the anterolateral thigh. Ultrasonography (US) is frequently used by physiatrists in the diagnosis and interventional treatment of musculoskeletal diseases. MP is usually diagnosed with clinical symptoms such as burning, tingling, pain, and dysesthesia in the anterolateral thigh. Electromyography, US, and magnetic resonance imaging are helpful in diagnosis. US is an easy-to-apply, inexpensive method in daily practice, providing great comfort to clinicians in determining etiology and differential diagnosis. Treatment may include patient education, avoiding tight belts, losing weight, conservative treatment methods, use of non-steroidal anti-inflammatory drugs, local anesthetic and/or steroid injections, surgical neurectomy, neurolysis or transpositions. However, in recent years, there have been case series showing that radiofrequency ablation (RF) can also be applied. The aim of this study is to compare the effectiveness of RF ablation of the lateral femoral cutaneous nerve with steroid injection in patients with clinically diagnosed MP and confirmed by US.

ELIGIBILITY:
Inclusion Criteria:

* Patients with numbness, tingling and pain in the anterolateral thigh region
* Patients with edematous LFCN observed on ultrasound and diagnosed with MP and with complaints resistant to conservative treatment
* Being literate

Exclusion Criteria:

* History of lumbar discopathy or history of discopathy surgery
* Cardiac pacemaker
* History of bilateral hip, knee, foot and lumbar region fractures
* History of previous hip and knee surgery
* Fixed joint contracture in the lower extremity
* History of malignancy and chemotherapy or radiotherapy
* Presence of any neuromuscular disease
* Progressive or non-progressive central and peripheral nervous system disease
* Patients in pregnancy and lactation
* Bleeding diathesis, INR>1.2
* Uncontrolled diabetes or other serious comorbidities
* Allergy to drugs or materials used
* Local infections or sepsis

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-11-01 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | Baseline, 1st day, 2nd week, 3rd month, 6th month
  The patients' pain levels were assessed using the Visual Analog Scale (VAS). The VAS pain score was scored as "no pain" (score=0) and "worst pain" (score=10).

SECONDARY OUTCOMES:
The Leeds Assessment of Neuropathic Symptoms and Signs pain scale | Baseline, 1st day, 2nd week, 3rd month, 6th month
  The Leeds Assessment of Neuropathic Symptoms and Signs pain scale will be used to assess the presence of neuropathic pain. It consists of two subcategories: pain questionnaire and sensory assessment. The questionnaire consists of five questions about general pain symptoms of the patient, and two questions, that are answered after appropriate clinical examination following predetermined methodology, which includes the seek for allodynia and altered pinprick threshold Scoring varies between 0 and 24 points, with a total score > 12 indicating pain predominantly of neuropathic etiology.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Merve Ata, MD, Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Mackinnon SE, Hudson AR, Gentili F, Kline DG, Hunter D. Peripheral nerve injection injury with steroid agents. Plast Reconstr Surg. 1982 Mar;69(3):482-90. doi: 10.1097/00006534-198203000-00014. PMID 7063571
- [Result] Ghai B, Dhiman D, Loganathan S. Extended duration pulsed radiofrequency for the management of refractory meralgia paresthetica: a series of five cases. Korean J Pain. 2018 Jul;31(3):215-220. doi: 10.3344/kjp.2018.31.3.215. Epub 2018 Jul 2. PMID 30013736
- [Result] Abd-Elsayed A, Gyorfi MJ, Ha SP. Lateral Femoral Cutaneous Nerve Radiofrequency Ablation for Long-term Control of Refractory Meralgia Paresthetica. Pain Med. 2020 Nov 7;21(7):1433-1436. doi: 10.1093/pm/pnz372. PMID 32022852
- [Result] Lee SH, Shin KJ, Gil YC, Ha TJ, Koh KS, Song WC. Anatomy of the lateral femoral cutaneous nerve relevant to clinical findings in meralgia paresthetica. Muscle Nerve. 2017 May;55(5):646-650. doi: 10.1002/mus.25382. Epub 2017 Jan 3. PMID 27543938